CLINICAL TRIAL: NCT01059331
Title: Perioperative Administration of Pregabalin in Laparoscopic Living Donor Nephrectomy (L-LDN) - an Adjuvance to Peroral Analgetic Treatment - a Randomized Controlled Study
Brief Title: Postoperative Analgesia After Laparoscopic Living Donor Nephrectomy
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Oslo University Hospital (Other)
Responsible Party: Principal Investigator, Marianne Myhre, cand.med., Oslo University Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2009/1286-1
Record Dates: First submitted 2010-01-28; First posted 2010-01-29 (Estimated); Last update posted 2014-03-21 (Estimated); Status verified 2014-03

CONDITIONS: Living Donors
Keywords: Kidney
MeSH Terms: interventions — Pregabalin; Sugars

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Pregabalin (Experimental)
  Interventions: Drug: Pregabalin
- Sugar pill (Placebo Comparator)
  Interventions: Drug: Sugar pill

INTERVENTIONS:
Drug: Pregabalin — 150 mg x 2 daily for 2 days
  Other Names: Lyrica ATC-nr.: NO3A X 160
  Arms: Pregabalin
Drug: Sugar pill — 1 tablet x 2 daily, for 2 days
  Arms: Sugar pill

SUMMARY:
The aim of the study is to investigate if perioperative administration of pregabalin vil reduce postoperative pain and the postoperative need for intravenous opioids compared with todays standard treatment which consist of paracetamol, corticoids and ketobemidone.

In addition potential sideeffects as sedation and effect on cognitive function will be recorded.

ELIGIBILITY:
Inclusion Criteria:

* >18, < 75 years
* healthy patients accepted for laparoscopic living donor nephrectomy

Exclusion Criteria:

* not familiar to the Norwegian language (spoken and written)
* allergic to one or more of the medication given in the study

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2010-02; Primary Completion 2011-10 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Opioid consumption in milligrams Pain Score given as Numeric Rating Scale (NRS) | Daily troughout the hospital stay, approx. 6 days

SECONDARY OUTCOMES:
Sedation and cognitive function | Daily troughout the hospital stay, approx. 6 days

CONTACTS AND LOCATIONS:
Overall Officials: Audun Stubhaug, dr.med., Principal Investigator — Universitetet i Oslo, Rikshospitaelt, Anestesi- og intensivavdelingen
Locations (1):
- Oslo Universitetssykehus, Rikshospitalet, Oslo, Norway

REFERENCES:
- [Background] Tiippana EM, Hamunen K, Kontinen VK, Kalso E. Do surgical patients benefit from perioperative gabapentin/pregabalin? A systematic review of efficacy and safety. Anesth Analg. 2007 Jun;104(6):1545-56, table of contents. doi: 10.1213/01.ane.0000261517.27532.80. PMID 17513656
- [Background] Mathiesen O, Jacobsen LS, Holm HE, Randall S, Adamiec-Malmstroem L, Graungaard BK, Holst PE, Hilsted KL, Dahl JB. Pregabalin and dexamethasone for postoperative pain control: a randomized controlled study in hip arthroplasty. Br J Anaesth. 2008 Oct;101(4):535-41. doi: 10.1093/bja/aen215. Epub 2008 Jul 23. PMID 18653493
- [Background] Agarwal A, Gautam S, Gupta D, Agarwal S, Singh PK, Singh U. Evaluation of a single preoperative dose of pregabalin for attenuation of postoperative pain after laparoscopic cholecystectomy. Br J Anaesth. 2008 Nov;101(5):700-4. doi: 10.1093/bja/aen244. Epub 2008 Aug 20. PMID 18716003
- [Background] Jokela R, Ahonen J, Tallgren M, Haanpaa M, Korttila K. A randomized controlled trial of perioperative administration of pregabalin for pain after laparoscopic hysterectomy. Pain. 2008 Jan;134(1-2):106-12. doi: 10.1016/j.pain.2007.04.002. Epub 2007 May 15. PMID 17507163
- [Background] Gilron I. Gabapentin and pregabalin for chronic neuropathic and early postsurgical pain: current evidence and future directions. Curr Opin Anaesthesiol. 2007 Oct;20(5):456-72. doi: 10.1097/ACO.0b013e3282effaa7. PMID 17873599